CLINICAL TRIAL: NCT00195221
Title: A Retrospective Study to Describe the Incidence of Moderate to Severe Allergic Reactions to Factor IX in Patients With Hemophilia B
Brief Title: Study to Describe the Allergic Reactions to Factor IX in Patients With Hemophilia B
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 3090A-101657
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Hemophilia B; Allergic Reactions
Keywords: Hemophilia B
MeSH Terms: conditions — Hemophilia B; Hypersensitivity

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Retrospective, multicenter study in patients with hemophilia B. This study will be placed at 20 to 50 hemophilia treatment centers in North America and the EU, and is designed to estimate the frequency of Class II and III allergic reactions in association with the administration of any FIX concentrate.

Following informed consent and eligibility, historical patient information including demographics, allergy history, hemophilia history, frequency and severity of allergic reaction(s), number of exposure days with products causing allergic reactions, exposure days to blood products including FIX concentrates, treatment for allergic reaction(s), outcome of event(s), any other adverse event(s) occuring within 48 hours of onset of allergic reaction(s), rechallenge and outcome, switch to another FIX product (if applicable) and outcome, current status of patient, and results of any special studies (eg, skin or RAST testing, alloantibody analyses, ect) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to release patient information
* Living or deceased patients with mild to severe hemophilia B who have had at least 1 exposure to replacement factor IX product(s).
* Living or deceased patients who had their first infusion of any FIX product between 1 January 1991 and 31 December 2003.

Exclusion Criteria:

* There are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166
Dates: Start 2005-02; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, MedInfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Austria, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For UK, ukmedinfo@wyeth.com; Trial Manager, Principal Investigator — For Italy, decresg@wyeth.com
Locations (38):
- United States (15):
  - Phoenix, Arizona
  - Orange, California
  - Atlanta, Georgia
  - Boise, Idaho
  - Peoria, Illinois
  - Iowa City, Iowa
  - East Lansing, Michigan
  - Rochester, Minnesota
  - New Brunswick, New Jersey
  - Dayton, Ohio
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Fort Worth, Texas
  - San Antonio, Texas
  - Seattle, Washington
- Vienna, Austria
- Belgium (2):
  - Brussels
  - Montegnée
- Calgary, Alberta, Canada
- France (4):
  - Liffré
  - Montmorency
  - Paris
  - Strasbourg
- Germany (2):
  - Hamburg
  - Münster
- Italy (9):
  - Catania
  - Catanzaro
  - Milan
  - Naples
  - Padua
  - Palermo
  - Parma
  - Perugia
  - Vicenza
- Spain (2):
  - Valencia
  - Valladolid
- United Kingdom (2):
  - Wolverhampton, Wstmid
  - Cardiff